CLINICAL TRIAL: NCT02731365
Title: Concurrent Deep Brain Stimulation (DBS) Local Field Potential Analysis and Stimulation in a Closed-Loop Neuromodulation Device
Brief Title: Concurrent DBS Local Field Potential Analysis and Stimulation in a Closed-Loop Neuromodulation Device
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped to await new generation of device anticipated to be released 2018.
Sponsor: Vibhor Krishna (Other)
Responsible Party: Sponsor-Investigator, Vibhor Krishna, Assistant Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014H0423
Record Dates: First submitted 2015-10-13; First posted 2016-04-07 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DBS LFP Activa PC+S (Experimental): The study aims at testing a slightly modified device (battery) that is similar to the approved system that has the potential of offering future patients a closed loop system with automatic adjustments of stimulation. The purpose of this clinical study is to allow the investigation of local field potential (LFP) signals in patients treated with DBS of the STN. This study will identify common LFP biomarkers observed as a function of disease symptoms, medication effect, fluctuations in disease, and changes resulting from adjustments from current standard practices of DBS programming.
  Interventions: Device: Activa PC+S

INTERVENTIONS:
Device: Activa PC+S — The Activa PC+S is a newly developed Medtronic DBS implantable system and is available for use in clinical research. This system has a mechanism for both sensing of LFP and the ability to provide deep brain stimulation therapy. The sensing capabilities are controllable with data management using a clinician sensing tablet programmer that has a USB extension allowing for telemetry to an encrypted, locked computer.

SUMMARY:
The purpose of this clinical study is to allow the investigation of local field potential (LFP) signals in patients treated with DBS of the STN. This study will identify common LFP biomarkers observed as a function of disease symptoms, medication effect, fluctuations in disease, and changes resulting from adjustments from current standard practices of DBS programming. The data collected and LFP markers identified will serve as guidelines for future stimulation predicted programming.

DETAILED DESCRIPTION:
The goals of this study are to evaluate local field potentials (LFP) and associated beta, gamma and other band oscillations and their correlation with disease pathophysiology and clinical status of the patients, and to potentially determine a more objective biomarker of response to deep brain stimulation (DBS) treatment. This study aims to find evidence that changes in the power and coherence of the beta and gamma bands can be consistently linked to DBS adjustment and associated clinical effects. This approach can be of significant potential benefit to provide a foundation for closed loop DBS therapy in patients with continuous DBS adjustments.

This study will use a novel bi-directional neural interface system that can chronically and simultaneously record, sense, process and telemeter LFP signals from DBS electrode (Rouse et al. 2011) to study the stability and subsequent change to LFP linked to the clinical state relevant to the present disorder, and DBS stimulation at rest and during motor and cognitive tasks. This investigation will be conducted at the Ohio State University.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are candidates for DBS surgery.
* Age 22-90 years of age
* Participant is willing to comply with all follow-up evaluations at the specified study time points.
* Participant is able to provide informed consent prior to enrollment in the study.
* The participant is fluent in English.

Exclusion Criteria:

* Significant cognitive impairment or dementia.
* Uncontrolled depression, anxiety or other mood disorder.
* Medical contraindications for general anesthesia, craniotomy, or DBS surgery.
* Diagnosis of acute myocardial infarction or cardiac arrest within previous 6 months.
* Condition requiring diathermy after DBS implantation.
* Subjects with any type of destruction and/or damage to the STN as determined by brain imaging.
* Co-morbid conditions that would interfere with study activities or response to treatment, which may include:
* Life expectancy < 3 years
* Severe Chronic pulmonary disease
* Intractable seizure disorders
* Local, systemic acute or chronic infectious illness
* Life threatening cardiac arrhythmias
* Severe collagen vascular disorder
* Kidney failure or other major organ systems failures
* History of a neurological ablation procedure.
* Labeled contraindication for MRI.
* History of hemorrhagic stroke.
* History of HIV infection or ongoing chronic infection (such as tuberculosis). Participation in another FDA device or medication trial that would interfere with the current study.

Ages: 22 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Identify and record LFP | 18 months
  The association between local field potential (LFP) signals in individuals who have undergone deep brain stimulation (DBS) of the subthalamic nucleus (STN) and successful completion of a cursor drive motor task.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Rezai, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center - Center for Neuromodulation, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No